CLINICAL TRIAL: NCT06672393
Title: A Multi-Center, Randomized, Double Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of HS-10374 in Adult Subjects With Moderate To Severe Plaque Psoriasis
Brief Title: A Study to Confirm Efficacy and Safety of HS-10374 for Moderate to Severe Plaque Psoriasis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10374-301
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-10374 (Experimental): Subjects will receive HS-10374 from Week 0 through Week 52.
  Interventions: Drug: HS-10374 6mg tablets
- Placebo (Placebo Comparator): Subjects will receive HS-10374 matching placebo from Week 0 through Week 16, and HS-10374 from Week 16 through Week 52.
  Interventions: Drug: HS-10374 6mg tablets; Drug: HS-10374-matched placebo tablets

INTERVENTIONS:
Drug: HS-10374 6mg tablets — Specified dose of HS-10374 tablets administered orally QD on specified days
Drug: HS-10374-matched placebo tablets — Specified dose of HS-10374-matched placebo tablets administered orally QD on specified days
  Arms: Placebo

SUMMARY:
This study has been designed to confirm the clinical efficacy and safety of HS-10374 in the treatment of moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a 52-week, multi-center, randomized, double-blind, placebo-controlled, Phase 3 study. The study duration includes a 4-week screening period, a 16-week placebo-controlled treatment period, a 36-week study drug treatment period, and a 4-week follow-up period. All eligible subjects will be randomly assigned in a 2:1 ratio to receive HS-10374 or placebo QD. At Week 16, subjects receiving placebo will be switched to HS-10374 QD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 years and older
* Diagnosis of plaque psoriasis for at least 6 months
* Eligible for phototherapy or systemic therapy
* Plaque covering ≥ 10% of BSA
* PASI ≥ 12, sPGA ≥3

Exclusion Criteria:

* Diagnosis of non-plaque psoriasis or drug-induced psoriasis
* Recent history of infection, history or risk of serious infection
* Any major illness or evidence of unstable condition of major organ systems including psychiatric disease
* Any condition possibly affecting the PK process of the study drug
* Evidence of other skin conditions that would interfere with the evaluation of psoriasis
* History of hypersensitivity to the ingredients of study drugs, history of anaphylaxis
* Prior exposure to TYK2 inhibitors
* Have received the prohibited treatment during the protocol required washout period
* Any significant laboratory or procedure abnormalities that might place the subject at unacceptable risk during this study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2025-10-22 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving PASI 75 response at Week 16 | Baseline to Week 16
  Psoriasis Area and Severity Index (PASI) is a scoring system quantifying the severity of psoriasis based on both lesion severity and area of involvement. PASI assessment is performed by investigators, and the numeric score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 75 response is defined as 75% or greater improvement in PASI score from baseline.
Proportion of patients achieving sPGA 0/1 with at least 2 points improvement from baseline at Week 16 | Baseline to Week 16
  Static physician's global assessment (sPGA) of psoriasis is an average assessment of all psoriatic lesions based on erythema, induration, and scale. It's a 5-point scale performed by investigators. A sPGA score of 0 or 1 means "clear" or "almost clear" respectively.

SECONDARY OUTCOMES:
Incidence, severity and association with the study drug of adverse events (AEs), serious AEs (SAEs), and AEs leading to discontinuation | Baseline to Week 56
Number of participants with clinical laboratory abnormalities | Baseline to Week 56
  Clinical laboratory tests include hematology, coagulation testing, blood chemistry, urinalysis, stool analysis, high-sensitivity C-reactive protein, etc.
Incidence of clinically significant changes in electrocardiogram (ECG) | Baseline to Week 56
  ECG parameters include heart rate, PR interval, RR interval, QRS duration, QTcF interval.
Number of participants with abnormalities of physical examination | Baseline to Week 56
  Physical examination includes assessments of general appearance, skin, lymph nodes, head, neck, lung, heart, abdomen, spine, extremities, nervous system, etc.
Number of participants with abnormalities of vital signs | Baseline to Week 56
  Vital signs measured include blood pressure, pulse rate, and temperature.
PASI 75 response rates at specified time points | Baseline to Week 56
  Psoriasis Area and Severity Index (PASI) is a scoring system quantifying the severity of psoriasis based on both lesion severity and area of involvement. PASI assessment is performed by investigators, and the numeric score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 75 response is defined as 75% or greater improvement in PASI score from baseline.
PASI 90 response rates at specified time points | Baseline to Week 56
  Psoriasis Area and Severity Index (PASI) is a scoring system quantifying the severity of psoriasis based on both lesion severity and area of involvement. PASI assessment is performed by investigators, and the numeric score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 90 response is defined as 90% or greater improvement in PASI score from baseline.
PASI 100 response rates at specified time points | Baseline to Week 56
  Psoriasis Area and Severity Index (PASI) is a scoring system quantifying the severity of psoriasis based on both lesion severity and area of involvement. PASI assessment is performed by investigators, and the numeric score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 100 response is defined as 100% improvement in PASI score from baseline.
Proportion of patients with sPGA 0/1 at specified time points | Baseline to Week 56
  Static physician's global assessment (sPGA) of psoriasis is an average assessment of all psoriatic lesions based on erythema, induration, and scale. It's a 5-point scale performed by investigators. A sPGA score of 0 or 1 means "clear" or "almost clear" respectively.
Proportion of patients with sPGA 0 at specified time points | Baseline to Week 56
  Static physician's global assessment (sPGA) of psoriasis is an average assessment of all psoriatic lesions based on erythema, induration, and scale. It's a 5-point scale performed by investigators. A sPGA score of 0 means "clear".
Proportion of patients achieving PSSD symptom score of 0 at specified time points among patients with a baseline symptom score ≥1 | Baseline to Week 56
  Psoriasis symptoms and signs diary (PSSD) is an 11-item patient-reported instrument. It assesses severity of 5 symptoms (itch, pain, stinging, burning, skin tightness) and 6 subject-observed signs (skin dryness, cracking, scaling, shedding or flaking, redness, bleeding). The severity of each item is rated from 0 (absent) to 10 (worst imaginable). Two subscores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Proportion of patients achieving DLQI 0/1 at specified time points among patients with a baseline DLQI score ≥2 | Baseline to Week 56
  The dermatology life quality index (DLQI) is a patient reported outcome measurement. It's a questionnaire consisting of 10 questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week. Each question is scored on a scale of 0 to 3, and the sum of each scores range from 0 (no impairment of life quality) to 30 (maximum impairment).
Proportion of patients achieving ss-PGA 0/1 at Week 16 among patients with a baseline ss-PGA score ≥3 | Baseline to Week 16
  Scalp specific physician's global assessment (sPGA) of psoriasis is an assessment of the disease severity of scalp psoriasis based on erythema, thickness, and scale. It's a 5-point scale performed by investigators. A sPGA score of 0 or 1 means "absence of disease" or "very mild disease" respectively.
Proportion of patients achieving PGA-F 0/1 at Week 16 among patients with a baseline PGA-F score ≥3 | Baseline to Week 16
  Physician's global assessment of fingernails (PGA-F) is a scale used to assess a patient's fingernail psoriasis. Ten fingernails on the hand will be globally evaluated separately for nail bed and nail matrix disease on a scale of 0 to 4. The overall global assessment of nails is the worse of the nail bed and nail matrix assessment. A PGA-F score of 0 or 1 means "clear" or "minimal" respectively.
Proportion of patients achieving pp-PGA 0/1 at Week 16 among patients with a baseline pp-PGA score ≥3 | Baseline to Week 16
  Palmoplantar PGA (pp-PGA) is a scale performed by investigators to assess a patient's palmoplantar psoriasis lesions on a scale of 0 to 4. A pp-PGA score of 0 or 1 means "clear" or "almost clear" respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China